CLINICAL TRIAL: NCT01063907
Title: An Open Label, Dose Escalation, Multicenter Phase 1/2 Study of KW-2478 in Combination With Bortezomib in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of KW-2478 in Combination With Bortezomib in Subjects With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2478-INT-001; 2009-016223-56 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: Leukemia; Immunoproliferative Disorder; Neoplasma by Histologic Type; Immune System Diseases; Hematologic Diseases; Blood Protein Disorders; Paraproteinemias; Multiple Myeloma; Hematologic Disorders; Leukemia, Chronic, B-cell; Leukemia, B-cell; Leukemia, Chronic; Neoplasms, Plasma Cell; Monoclonal Gammopathy of unknown significance (MGUS)
MeSH Terms: conditions — Multiple Myeloma; Leukemia; Immunoproliferative Disorders; Immune System Diseases; Hematologic Diseases; Blood Protein Disorders; Paraproteinemias; Leukemia, B-Cell; Bronchiolitis Obliterans Syndrome; Neoplasms, Plasma Cell; Monoclonal Gammopathy of Undetermined Significance | interventions — KW-2478; Hsp90 inhibitor KU757; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase 1: Cohort 1 (Experimental): Cohort 1: KW 2478 130 mg/m^2 and Bortezomib 1.0 mg/m^2
  Interventions: Drug: KW-2478; Drug: Bortezomib
- Phase 1: Cohort 2 (Experimental): Cohort 2: KW 2478 130 mg/m^2 and Bortezomib 1.3 mg/m^2
  Interventions: Drug: KW-2478; Drug: Bortezomib
- Phase 1: Cohort 3 (Experimental): Cohort 3: KW 2478 175 mg/m^2 and Bortezomib 1.0 mg/m^2
  Interventions: Drug: KW-2478; Drug: Bortezomib
- Phase 1: Cohort 4 (Experimental): Cohort 4: KW 2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2
  Interventions: Drug: KW-2478; Drug: Bortezomib
- Phase 2 (Experimental): KW 2478 175 mg/m^2 and Bortezomib 1.0 mg/m^2
  Interventions: Drug: KW-2478; Drug: Bortezomib

INTERVENTIONS:
Drug: KW-2478 — Administered Days 1, 4, 8 and 11 of a 21 day cycle
  Other Names: HSP90 Inhibitor
Drug: Bortezomib — Administered on Days 1, 4, 8 and 11 of a 21 day cycle
  Other Names: Velcade

SUMMARY:
The purpose of this study is to assess the safety and benefits of the investigational study drug, KW-2478, when given with bortezomib (Velcade®), a drug approved for the treatment of Multiple Myeloma (MM).

The primary objectives:

* To establish the safety, tolerability, and recommended Phase II dose (RP2D) of KW-2478 in combination with bortezomib (Phase I);
* To assess the overall response rate (ORR) when subjects with advanced MM are treated (Phase II).

The secondary objectives:

* To characterize the Pharmacokinetic (PK) and Pharmacodynamic (PD) of KW-2478 with bortezomib (Phase I only);
* To evaluate for preliminary evidence of efficacy (Phase I);
* To determine progression free survival (PFS) and duration of response of KW-2478 with bortezomib (Phase II).

DETAILED DESCRIPTION:
This is a multicenter, open label, dose escalation, Phase I / II study in subjects with relapsed and/or refractory MM. Up to 24 subjects to be enrolled in the Phase I to determine the RP2D. Up to 77 additional evaluable subjects to be enrolled in Phase II for a maximum up to 101 subjects treated in the study. Study centers in the USA and the UK will participate in Phase I and II. Centers in the Philippines will be participating in Phase II only. The planned enrollment period is 22 months and the planned study duration is 28 months.

ELIGIBILITY:
Accepts Healthy Volunteers: No

Inclusion Criteria:

1. Subjects with a confirmed diagnosis of Multiple Myeloma who have had one and no more than three prior regimens for MM to which they did not respond (failed) or from which they have relapsed.
2. Signed either an IRB or IEC approved informed consent
3. ECOG performance status of ≤ 2
4. Life expectancy of at least 3 months
5. M protein in either serum or urine, or free light chains if not measurable M protein in serum or urine, and clonal bone marrow plasma cells > 10%, and evidence of end organ damage
6. Adequate hematologic status, liver and renal function
7. Subjects of reproductive potential must agree to follow accepted pregnancy prevention methods during the study.

Exclusion Criteria:

1. No anti-cancer treatment for ≥ 4 weeks and no bortezomib treatment ≥ 60 days prior to receiving study drug
2. Any other severe, acute or chronic illness
3. No other prior or concurrent malignancy
4. No immunosuppressant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2010-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Kyowa Hakko Kirin Pharma, Inc.; Loan Hoang-Sayag, MD, Study Chair — Quintiles, Inc.; Noel Pingoy, MD, Study Chair — Gleneagles CRC
Locations (26):
- United States (9):
  - Arizona Clinical Research Center, Inc. / Arizona Oncology Associates, 1825 N Kolb,, Tucson, Arizona
  - Pacific Shores Medical Group 1043 Elm Ave, Suite 104, Long Beach, California
  - UCLA Medical Center Hematology / Oncology Division, 10945 Le Conte Ave #2333,, Los Angeles, California
  - Collaborative Research Group 2320 S Seacrest Blvd, Suite 202, Boynton Beach, Florida
  - Rush University Medical Center / Division of Hematology/Oncology Research 1725 W Harrison Street, Suite 834, Chicago, Illinois
  - Cancer Institute of New Jersey 195 Little Albany Street, New Brunswick, New Jersey
  - The Jones Clinic 7710 Wolf River Circle, Germantown, Tennessee
  - UT MD Anderson Cancer Center, 1515 Holcombe Boulevard,, Houston, Texas
  - Gundersen Clinic Center for Cancer and Blood Disorders, 1900 South Ave, EB2-001,, La Crosse, Wisconsin
- Philippines (4):
  - The Medical City, 1609 MATI Building, The Medical City, Ortigas Avenue,, Pasig, Manila
  - National Kidney and Transplant Institute, Rm 3215 Doctors Clinic, East Avenue, Diliman, Quezon City
  - Makati Medical Center, New Wing Hall C372, #2 Amorsolo Street, Legaspi Village,, Makati City
  - Saint Lukes Medical Center, Rm 222 MAB Saint Lukes Medical Center, E. Rodriguez, Quezon City
- United Kingdom (13):
  - Darent Valley Hospital Dept of Haematology, Acorn House, Darenth Wood Road, Dartford, Kent
  - St Bartholomew's Hospital Haematology Department, 1st Floor, Pathology, Barbican, London
  - Christie Hospital - Department Haematology, 550 Wilmslow Road, Withington, Manchester, Greater Manchester
  - Hillingdon Hospital Dept of Haematology, Pield Health Road, Uxbridge, Middlesex
  - Royal Marsden Hospital, Orchard House, Sutton, Surrey
  - Royal Bournemouth Hospital, Dept. of Haematolgy, Castle Lane East,, Bournemouth
  - Royal Devon & Exeter Hospital Haematology Centre, Barrack Road, Exeter
  - Northwick Park Hospital Dept of Haematology, Watford Road, Harrow
  - St James Hospital, St James' Institute of Oncology, Department of Haematology, Level 03, Bexley Wing,, Leeds
  - UCL Cancer Institute, Paul O'Gorman Building, University College London,72 Huntley Street, London
  - Manchester Royal Infirmary Dept of Haematology, Oxford Road, Manchester
  - Nottingham University Hospitals NHS Trust, Centre for Clinical Haemotology, Nottingham
  - Royal Cornwall Hospital Haematology Clinic, Truro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study centers in the USA and the UK participated in the Phase 1 portion, and study centers in the USA, UK, and Philippines participated in the Phase 2 portion.
Groups:
- Phase 1: KW-2478 and Bortezomib: The target population in Phase 1 were adults (≥18 years) of either gender with a confirmed history of MM by IMWG criteria had relapsed or failed to respond to 1-3 prior MM regimens with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 and a life expectancy ≥ 3 months. Subjects had to have disease that could be evaluated by serum or urinary levels of M protein or serum free light chains in the absence of measurable M protein in serum or urine.
  For Phase 1, the design was a standard 3+3 study of KW-2478 (130 or 175 mg/m^2) and bortezomib(1.0 or 1.3 mg/m^2) on Days 1, 4, 8, and 11 of a 21-day cycle utilizing four dose-escalation cohorts.
- Phase II: KW-2478 130mg/m^2 and Bortezomib 1.3mg/m^2: The target population in Phase 2 were adults (≥18 years) of either gender with a confirmed history of MM by IMWG criteria had relapsed or failed to respond to 1-3 prior MM regimens with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 and a life expectancy ≥ 3 months. Subjects had to have disease that could be evaluated by serum or urinary levels of M protein or serum free light chains in the absence of measurable M protein in serum or urine.
  For the Phase 2 portion of the study was designed to determine the preliminary efficacy of KW 2478 and bortezomib at the RP2D (KW-2478 175 mg/m^2/bortezomib1.3 mg/m^2).
Period: Overall Study
Arm/Group | Phase 1: KW-2478 and Bortezomib | Phase II: KW-2478 130mg/m^2 and Bortezomib 1.3mg/m^2
Started | 15 | 80
Completed | 15 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of up to 101 male and female subjects at least 18 years of age with a confirmed diagnosis of MM, who failed at least 1 and no more than 3 prior chemotherapy regimens and met other inclusion criteria and none of exclusion criteria, were to be enrolled in this study over a period of 22 months (up to 24 subject in P1 and 77 subjects in P2).
Groups:
- KW-2478 and Bortezomib: The target population in both Phase 1 and 2 were adults (≥18 years) of either gender with a confirmed history of MM by IMWG criteria had relapsed or failed to respond to 1-3 prior MM regimens with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 and a life expectancy ≥ 3 months. Subjects had to have disease that could be evaluated by serum or urinary levels of M protein or serum free light chains in the absence of measurable M protein in serum or urine.
  For Phase 1, the design was a standard 3+3 study of KW-2478 (130 or 175 mg/m^2) and Bortezomib(1.0 or 1.3 mg/m^2) on Days 1, 4, 8, and 11 of a 21-day cycle utilizing four dose-escalation cohorts (overall N=15). The Phase 2 portion of the study enrolled 80 subjects to determine the preliminary efficacy of KW 2478 and Bortezomib at the RP2D (KW-2478 175 mg/m^2 / Bortezomib 1.3 mg/m^2).
Arm/Group | KW-2478 and Bortezomib
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 61
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 18
  Philippines | 20
  United Kingdom | 57
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.87 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: To Establish the Safety, Tolerability, and RP2D (Phase 1); To Assess the Overall Response Rate in Subjects With Advanced Multiple Myeloma (Phase 2).
Description: The safety of KW-2478 was determined by reported TEAEs, observed DLTs, changes in PEs, vital sign measurements, ECGs, and laboratory analyses.
  The ORR, was defined as the best response over a specified number of cycles (calculated and summarized).
  Disease control rate (DCR) was defined as the best response over a specified number of cycles (calculated and summarized). Progression-free survival was defined as the time from the first day of treatment until the date of disease progression or death is first reported (calculated and summarized).
Time Frame: 21 day cycle, up to 52 weeks
Population: All subjects who received at least 1 dose, including a partial dose, of KW-2478 were evaluated for safety.
Measure: Number; unit: participants
Groups:
- Phase 1 & 2: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2: The target population in both Phase 1 and 2 were adults (≥18 years) of either gender with a confirmed history of MM by IMWG criteria had relapsed or failed to respond to 1-3 prior MM regimens with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 and a life expectancy ≥ 3 months. Subjects had to have disease that could be evaluated by serum or urinary levels of M protein or serum free light chains in the absence of measurable M protein in serum or urine.
  The Phase 1 portion of the study was a standard 3+3 study design of KW-2478 (130 or 175 mg/m^2) and Bortezomib (1.0 or 1.3 mg/m^2) on Days 1, 4, 8, and 11 of a 21-day cycle utilizing four dose-escalation cohorts.
  The Phase 2 portion of the study was designed to determine the preliminary efficacy of KW 2478 and Bortezomib at the RP2D (KW-2478 175 mg/m^2/Bortezomib 1.3 mg/m^2).
- Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0mg/m^2: Cohort 1: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle with a standard 3+3 study design.
- Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3mg/m^2: Cohort 2: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle with a standard 3+3 study design.
- Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0mg/m^2: Cohort 3: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle with a standard 3+3 study design.
- Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2: Cohort 4: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle with a standard 3+3 study design.
- Phase 2: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2: Phase 2: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle designed to determine the preliminary efficacy of KW 2478 and Bortezomib at the RP2D (KW-2478 175 mg/m^2/Bortezomib 1.3 mg/m^2).
Arm/Group | Phase 1 & 2: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2 | Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3mg/m^2 | Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2 | Phase 2: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2
Number analyzed (Participants) | 95 | 3 | 3 | 3 | 6 | 80
participants
  Subjects with Any TEAE | 95 | 3 | 3 | 3 | 6 | 80
  Related TEAE | 88 | 3 | 3 | 2 | 6 | 74
  Moderate (CTCAE 2) TEAE | 22 | 0 | 0 | 0 | 0 | 22
  Severe (CTCAE 3) TEAE | 54 | 3 | 2 | 2 | 5 | 42
  Life Threatening TEAE | 13 | 0 | 1 | 0 | 0 | 12
  Serious Treatment-Emergent AE | 48 | 2 | 3 | 3 | 4 | 36
  Subjects with Any DLT | 1 | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Phase 1: PK Absorption Tmax hr Day 11
Description: Descriptive summary statistics (number, arithmetic mean, standard deviation [SDev], coefficient of variation [CV%]) for concentration and PK data for KW-2478 and Bortezomib in Phase 1 were presented by cohort, dose level and day.
Time Frame: PK collected Day 11 of 21-day cycle
Population: The PK of KW-2478 was characterized after single administrations through @25 hours post start of infusion dose on Day 1 and through @7 hours post start of infusion dose on Day 11in Phase 1 only.
Measure: Mean (Standard Deviation); unit: hr
Groups:
- Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0mg/m^2; Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3mg/m^2; Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0mg/m^2; Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2: Both agents administered on Days 1, 4, 8 and 11 of a 21 day cycle
Arm/Group | Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3mg/m^2 | Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 6
hr | 1.03 (0.0441) | 1.03 (0.0481) | 1.11 (0.129) | 1.07 (0.0638)

3. Secondary Outcome: Phase 1: PK Exposure Cmax ng/mL Day 11
Description: as for outcome 2
Time Frame: PK collected Day 11 of 21-day cycle
Population: The PK of KW-2478 was characterized after single administrations through @25 hours post start of infusion dose on Day 1 and through @7 hours post start of infusion dose on Day 11 in Phase 1 only.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3mg/m^2 | Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 6
ng/mL | 7910 (5360) | 41000 (64100) | 5990 (2720) | 5280 (2290)

4. Secondary Outcome: Phase 1: PK Exposure AUC0-t hr*ng/mL Day 11
Description: as for outcome 2
Time Frame: PK collected Day 11 of 21-day cycle
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3mg/m^2 | Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 6
hr*ng/mL | 7940 (2580) | 26200 (36700) | 7190 (2150) | 6040 (2280)

5. Secondary Outcome: Phase 1: PK Elimination t½ hr Day 11
Description: as for outcome 2
Time Frame: PK collected Day 11 of 21-day cycle
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3mg/m^2 | Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0mg/m^2 | Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 6
hr | 1.88 (0.076) | 2.02 (0) | 1.84 (0.206) | 1.77 (0.262)

ADVERSE EVENTS:
Groups:
- Phase 1 and 2: KW-2478 and Bortezomib: KW-2478 and bortezomib: KW 2478 and bortezomib given on Days 1, 4, 8 and 11 of a 21 day cycle
- Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0 mg/m^2: Cohort 1: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle with a standard 3+3 study design.
- Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3 mg/m^2: Cohort 2: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle with a standard 3+3 study design.
- Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0 mg/m^2: Cohort 3: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle with a standard 3+3 study design.
- Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2: Cohort 4: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle with a standard 3+3 study design.
- Phase 2: KW-2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2: Phase 2: Both agents administered on Days 1, 4, 8, and 11 of a 21-day cycle designed to determine the preliminary efficacy of KW 2478 + BTZ at the RP2D (KW-2478 175 mg/m^2/BTZ 1.3 mg/m^2).
Arm/Group | Phase 1 and 2: KW-2478 and Bortezomib | Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0 mg/m^2 | Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3 mg/m^2 | Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0 mg/m^2 | Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2 | Phase 2: KW-2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2
Serious Adverse Events (participants affected / at risk) | 48/95 | 2/3 | 3/3 | 3/3 | 4/6 | 36/80
Other Adverse Events (participants affected / at risk) | 95/95 | 3/3 | 3/3 | 3/3 | 6/6 | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 and 2: KW-2478 and Bortezomib (N=95) | Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0 mg/m^2 (N=3) | Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3 mg/m^2 (N=3) | Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0 mg/m^2 (N=3) | Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2 (N=6) | Phase 2: KW-2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2 (N=80)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Listeriosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Troponin T increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 and 2: KW-2478 and Bortezomib (N=95) | Phase 1 Cohort 1: KW-2478 130 mg/m^2 and Bortezomib 1.0 mg/m^2 (N=3) | Phase 1 Cohort 2: KW-2478 130 mg/m^2 and Bortezomib 1.3 mg/m^2 (N=3) | Phase 1 Cohort 3: KW-2478 175 mg/m^2 and Bortezomib 1.0 mg/m^2 (N=3) | Phase 1 Cohort 4: KW-2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2 (N=6) | Phase 2: KW-2478 175 mg/m^2 and Bortezomib 1.3 mg/m^2 (N=80)
Anaemia (Blood and lymphatic system disorders) | 17 (30) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 14 (27)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 15 (37) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 14 (36)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (41) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 17 (39)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Erythema of eyelid (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye discharge (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Eye pruritus (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelids pruritus (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Foreign body sensation in eyes (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lacrimation increased (Eye disorders) | 12 (15) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 8 (10)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metamorphopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Retinal disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 16 (19) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 12 (15)
Visual acuity reduced (Eye disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 13 (19) | 2 (6) | 0 (0) | 2 (2) | 0 (0) | 9 (11)
Abdominal pain (Gastrointestinal disorders) | 17 (31) | 2 (5) | 0 (0) | 1 (1) | 1 (4) | 13 (21)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 11 (12) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 42 (71) | 3 (8) | 2 (4) | 2 (2) | 2 (3) | 33 (54)
Diarrhoea (Gastrointestinal disorders) | 70 (199) | 3 (29) | 2 (9) | 3 (7) | 4 (6) | 58 (148)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 13 (20) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 10 (16)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (5) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 55 (114) | 3 (11) | 1 (2) | 1 (2) | 5 (6) | 45 (93)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 38 (72) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 35 (67)
Asthenia (General disorders) | 15 (17) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 13 (15)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Chest pain (General disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Chills (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 51 (101) | 2 (6) | 3 (10) | 2 (2) | 3 (4) | 41 (79)
Feeling cold (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Infusion related reaction (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infusion site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 12 (17) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 9 (12)
Pain (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 12 (15) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 10 (11)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 14 (19) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 11 (14)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Rhinitis (Infections and infestations) | 7 (13) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 6 (10)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 14 (15) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 13 (14)
Urinary tract infection (Infections and infestations) | 6 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Viral infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Narcotic intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Blood magnesium decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood potassium decreased (Investigations) | 4 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (11) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (10)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Protein total increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 9 (10) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 7 (7)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 28 (44) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 25 (38)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid intake reduced (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (13) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (10)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 10 (11)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dactylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (13)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (17) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 10 (15)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (19) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 13 (17)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Areflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 25 (33) | 3 (8) | 0 (0) | 1 (1) | 3 (3) | 18 (21)
Dizziness exertional (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 13 (13) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 10 (10)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 23 (41) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 20 (38)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperreflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 8 (11) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 5 (7)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyporeflexia (Nervous system disorders) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 8 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (13)
Neuropathy peripheral (Nervous system disorders) | 28 (48) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 24 (42)
Paraesthesia (Nervous system disorders) | 11 (17) | 0 (0) | 2 (5) | 1 (2) | 1 (1) | 7 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (36) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 14 (35)
Presyncope (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Sensory loss (Nervous system disorders) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 13 (15) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 10 (12)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (29) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 16 (23)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (25) | 2 (2) | 1 (5) | 2 (2) | 1 (2) | 13 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 9 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 13 (17) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 11 (12)
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 5 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9)
Orthostatic hypotension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Phlebitis (Vascular disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Thrombophlebitis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vasculitis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vein discolouration (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less